CLINICAL TRIAL: NCT04731376
Title: Perioperative Testosterone Replacement Therapy Improves Outcomes: A Pilot Safety and Feasibility Study
Brief Title: Perioperative Testosterone Replacement Therapy for the Improvement of Post-Operative Outcomes in Patients With Low Testosterone
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenneth Ogan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001062; NCI-2020-06998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU5097-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-02-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hypogonadism; Malignant Urinary System Neoplasm; Urinary System Disorder; Urinary System Neoplasm
MeSH Terms: conditions — Hypogonadism; Urologic Neoplasms; Urologic Diseases | interventions — Practice Guidelines as Topic; Standard of Care; testosterone 17 beta-cypionate; Testosterone Propionate; Methyltestosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (testosterone cypionate) (Experimental): Patients with low testosterone levels receive testosterone cypionate IM QW for 3 months.
  Interventions: Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate
- Arm II (best practice) (Active Comparator): Patients with normal testosterone levels receive standard peri-operative care.
  Interventions: Other: Best Practice; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard peri-operative care
  Other Names: standard of care; standard therapy
  Arms: Arm II (best practice)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies; Quality of life questionnaires will be given both preoperatively and at 3-months postoperatively
Drug: Testosterone Cypionate — Given IM
  Other Names: depAndro; Depo-Testosterone; Depotest; Depovirin; Pertestis; Virilon
  Arms: Arm I (testosterone cypionate)

SUMMARY:
This phase I trial investigates the safety of testosterone replacement therapy around the time of major urologic surgery (perioperative) in order to improve quality of life and post-operative outcomes such as decreased length of hospital stay, complications, and mortality in patients with low testosterone levels. Studies have demonstrated that patients undergoing testosterone replacement therapy have increased lean body mass, decreased fat mass and have improved physical function. Testosterone replacement therapy can also stimulate bone formation and may decrease the risk of fracture. Information from this trial may be used to support the incorporation of testosterone level testing and testosterone replacement into the perioperative treatment decision-making process.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the safety and feasibility of perioperative testosterone replacement (TR) therapy in hypogonadal male patients undergoing major operations.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients with low testosterone levels receive testosterone cypionate intramuscularly (IM) once a week (QW) for 3 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients with normal testosterone levels receive standard peri-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled for major surgery requiring an overnight hospital stay
* Patients must be able to give informed consent
* Patients must be willing to do study's preoperative and post-operative assessment tools

Exclusion Criteria:

* Patient with history of prostatectomy with detectable prostate specific antigen (PSA)
* Patient with history of prostate radiation/chemotherapy treatment and has experienced bounce or rise in PSA
* Patients with history of/undergoing orchiectomy
* Patients undergoing hormone replacement therapy currently or history of testosterone use within last year
* Patients who use anabolic steroids
* Patients with history of solitary or undescended testis
* Patients with history of pituitary disorders
* Patients with history of thromboembolic events in last year
* Patients with hematocrit > 55%
* Patients with uncontrolled congestive heart failure
* Special populations: Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women and prisoners

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life before and after surgery | Baseline to 3 months
  The Patient Reported Outcomes Measurement Information System (PROMIS Global Health-10) is a 10 question survey that uses questions concerning physical function, overall quality of life, physical health, mood, ability to participate in social roles and activities, pain and fatigue to arrive at a score between 10 and 50. Patient's score are the outcome we will measure.
Change in frailty phenotype before and after surgery | Baseline, post operative refers to the period after the procedure until final follow up and study completion. Will occur an average of 90 days after the procedure.
  The Fried Frailty Criteria uses a comorbidity scale, measures of activity, physical tests of strength and speed, nutritional status and anatomic features to produce a score from 0-5. These numbers correspond with the following frailty categorizations: non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5). This score represents one outcome measure.
Major complications | Within 90 days of surgery
  Major complication considered Clavien-Dindo IIIb and above.
Minor complications | Within 90 days of surgery
  Minor complication considered Clavien-Dindo IIIb and below.
Rate of intensive care unit (ICU) admission | Up to 3 months post-surgery
  Admissions to the ICU between post-op day 1 to 90 days post surgery
Hospital length of stay | Up to 3 months post-operative
  Number of days stayed in the hospital after surgery
Discharge disposition | Discharge from hospital
  Determined by if patient is discharged to home, to home with services, or to facility.
Unplanned readmissions | Within 90 days of surgery
  Readmissions to hospital after discharge within 90 days
Mortality rate | Within 90 days of surgery
  Rate of patient deaths after surgery
Testosterone level | Up to 3 months post-operative
  Levels of Testosterone determined by laboratory blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States